CLINICAL TRIAL: NCT04922372
Title: Surface Texture and Clinical Performance of Milled BioHPP Polyetheretherketone (PEEK) Single Posterior Crowns Veneered With Two Different Techniques (Randomized Controlled Clinical Trial)
Brief Title: Surface Texture and Clinical Performance of Milled BioHPP Polyetheretherketone (PEEK) Single Posterior Crowns Veneered With Two Different Techniques
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Kamal Ibrahim Hassan, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 261020
Record Dates: First submitted 2021-06-05; First posted 2021-06-10 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Surface Roughness
MeSH Terms: interventions — polyetheretherketone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm copping veneered with composite resin (Experimental)
  Interventions: Combination Product: peek
- control arm copping veneered with manual layering (Active Comparator)
  Interventions: Combination Product: peek

INTERVENTIONS:
Combination Product: peek — After tooth preparation, adequate 2ry Impression using non aqueous elastomeric impression materials and bite registration will be taken. 5. Fabrication of the temporary restoration using composite resin temporary material and cemented using non Eugenol Zinc Oxide temporary cement. 11.a.iii. Fabrication and cementation of restoration: Bio-HPP will be supplied in the form of discs to fabricate crown core by CAD/CAM technology then veneered with two veneering techniques; the CAD/ CAM and the manual technique using the visio.lign system of appropriate shade. The finished Bio HPP crown will be cemented by adhesive resin cement according to manufacturer instruction

SUMMARY:
Research question:

For patients requiring posterior single crowns, does the use of Milled BioHPP PEEK copings veneered with CAD/CAM composite resin offer better surface texture and clinical performance when compared Milled BioHPP PEEK copings veneered with manual layering?

Statement of the problem Nowadays, metal free restorations are widely used. PEEK is one among these restorations that has many applications in dental field. Owing to PEEK's excellent mechanical properties, it is gaining popularity in prosthodontics. The opaque nature of PEEK allows its use as a framework material in fixed prosthodontics and composite resin material is used as a veneering material to achieve aesthetics .

The compatible composite veneering material can be manufactured by both manual and CAD/CAM techniques. Yet, there is no enough research regarding the influence of the veneering technique on the surface texture and clinical performance of these restorations.

Rationale PEEK combination of mechanical properties and high biocompatibility make it a very promising material . PEEK based crowns are veneered by composite resin material. Among the methods of fabrication of veneering composite is the manual layering and CAD/CAM techniques . The surface flaws and internal defects determine the strength of the material and affects its performance . Accordingly the evaluation of the veneering technique is mandatory.

The rationale for carrying out this study lies in providing an alternative solution to the manual veneering technique, which will, in-turn, provide better surface properties and clinical performance of the restoration and accordingly increase its longevity.

Aim of the study:

- The aim of this study is to evaluate the surface texture and clinical performance of milled BioHPP PEEK veneered with CAD/CAM composite resin and compare them to milled BioHPP PEEK veneered manually.

Null hypothesis:

There is no difference in the surface texture and clinical performance between milled BioHPP PEEK veneered with CAD/CAM composite resin and milled BioHPP PEEK veneered manually.

Primary objective:

* Primary outcome: (surface texture) of the two groups will be assessed using the modified USPHS.
* Secondary outcome: (fracture) of the two groups will be assessed using the modified Ryge criteria.

DETAILED DESCRIPTION:
Intervention: Examination and diagnosis: - Selection and examination of the patients according to inclusion and exclusion criteria. Diagnosis of the patients' chief complaint and teeth that will be involved in this study will be done then performing proper scaling and polishing procedure, Primary impression will be taken to produce study cast. The patients will be asked to maintain good oral hygiene measures by using tooth brush twice daily. - Taking a pre-operative professional photo, Tooth preparation procedure: Recording the sulcus depth and gingival condition prior to preparation, Conservative tooth preparation will be prepared after local anesthesia has been given as required., Full coverage preparation will be carried out , After tooth preparation, adequate 2ry Impression using non aqueous elastomeric impression materials and bite registration will be taken., Fabrication of the temporary restoration using composite resin temporary material and cemented using non Eugenol Zinc Oxide temporary cement, Fabrication and cementation of restoration: Bio-HPP will be supplied in the form of discs to fabricate crown core by CAD/CAM technology then veneered with two veneering techniques; the CAD/ CAM and the manual technique using the visio.lign system of appropriate shade. The finished Bio HPP crown will be cemented by adhesive resin cement according to manufacturer instruction, Criteria for discontinuing: Restoration will be removed when there are any signs of leakage, fracture or severe post-operative pain due to pulpal response and replaced by a temporary restoration cemented with Ca (OH) cement in order to alleviate pain, Strategies to improve adherence to intervention protocol: - ''In the first visit, a Face to Face adherence session will be held in which the patient should be informed about the study steps and how to maintain oral hygiene measures. Further sessions will occur at the follow-up visits.8 Participant patients will be asked about any problems they are having. Patients will be recalled every three months for one year for follow up visits. Permitted or prohibited interventions: Oral hygiene measures are permitted for enhanced results while using hard tooth brushes or abrasive containing tooth paste after intervention are prohibited

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

All subjects are required to be:

1. From 18-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations.
3. Psychologically and physically able to withstand conventional dental procedures.
4. Patients in a need for posterior crown.
5. Able to return for follow-up examinations and evaluation Exclusion criteria 1. Patient less than 18 or more than 50 years 2. Patient with active resistant periodontal diseases 3. Patients with poor oral hygiene and uncooperative patients 4. Pregnant women 5. Patients in the growth stage with partially erupted teeth 6. Psychiatric problems or unrealistic expectations 7. Lack of opposing dentition in the area of interest.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-07-22 (Estimated); Primary Completion 2022-07-22 (Estimated); Study Completion 2022-12-22 (Estimated)

PRIMARY OUTCOMES:
surface texture | one year
  Alpha: Surface is smooth as the surrounding, Bravo: Surface is rough than the surrounding, Charlie: Surface is very rough avoiding movement of the explorer, Delta: New restoration is needed.

SECONDARY OUTCOMES:
fracture | one year
  Alpha: Smooth surface of the restoration (shiny after air drying) Bravo: Dull surface and/or chipping of veneering material that does not impair function Charlie: Chipping of veneering material impairing esthetics and function and/or exposing framework material

IPD SHARING:
Plan to Share IPD: Yes
The patient will be treated in visits designated as follows:
  * Visit 1: Preoperative records, face-to-face adherence reminder session, clinical, radiographic examination, intraoral photographs and primary impression (alginate impression*) for diagnostic cast construction.
  * Visit 2: Teeth preparation, secondary impression using addition silicone rubber base material and temporary restoration.
  * Visit 3: placement and temporary cementation of the interim restoration using temporary cement.
  * Visit 4: try in of the coping.
  * Visit 5: placement of final restoration. Evaluation of the restoration immediately and follow up visit every 3 months at (T0, T6, T12)